CLINICAL TRIAL: NCT02047721
Title: The Effects of Exercise on Appetite Regulation in Overweight/Obese Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13-3252; UL1TR001082 (NIH)
Record Dates: First submitted 2014-01-15; First posted 2014-01-28 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Exercise; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Intervention (Experimental): A supervised exercise program
  Interventions: Behavioral: Exercise
- Nutritional Intervention (Experimental): A supervised diet program
  Interventions: Behavioral: Diet

INTERVENTIONS:
Behavioral: Exercise — The intervention gradually increases EE from 150-200 kcal/day 5 days per week to a target of 400 kcal/d 5 days per week and will last a total of 12 weeks.
  Arms: Physical Intervention
Behavioral: Diet — A supervised diet program which has been successfully implemented by our group with a goal being to reduce energy intake by ~2000 kcal/week.
  Arms: Nutritional Intervention

SUMMARY:
In this study the Investigators are examining the effects of a 12-week exercise program (intervention) on measures of appetite and food intake regulation in overweight to mildly obese healthy adults. The Investigators hypothesize that individuals who lose a significant amount of weight in response to the intervention will show a reduction in the brain response to food cues as measured by functional magnetic resonance imaging (fMRI) when compared to those who do not lose weight. These changes in neuronal activity will be associated to physiologic and behavioral measures.

ELIGIBILITY:
Inclusion Criteria:

* all ethnic groups and both genders;
* age: 21-45 yrs;
* BMI: 27-35;
* weight stable within +/- 5 percent in the last 6 months;
* sedentary (less than 1 hour of planned physical activity by self-report).

Exclusion Criteria:

* history of cardiovascular disease (CVD), diabetes mellitus, uncontrolled hypertension, untreated thyroid disease, renal disease, hepatic disease, or any other medical condition affecting weight or energy metabolism;
* unable to effectively exercise due to cardiac, pulmonary, neurologic or orthopedic reasons;
* unable to pass screening graded exercise treadmill test;
* currently smoking;
* medications affecting weight, Energy Intake (EI) or Energy Expenditure (EE) in the last 6 months;
* weight loss or weight gain of >5 percent in past 6 months;
* currently pregnant, lactating or less than 6 months post-partum;
* bariatric surgery;
* major psychiatric disorder, presence of alcohol or substance abuse, current depression by history and/or a score >21 on the he Center for Epidemiologic Studies Depression Scale (CES-D), history of eating disorders and/or a score of >20 on the EATS-26;
* contraindication to MRI

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2014-02; Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
fMRI Response to Visual Food Cues | 12 weeks
  The neuronal response will be assessed by functional magnetic resonance imaging (fMRI) in response to visual food cues
  Blood oxygen dependent signal (BOLD) response in exposure to visual food cues will be measured during a fMRI scan and the difference between responses in those who lose weight vs. those who do not lose weight will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Legget, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Univeristy of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No